CLINICAL TRIAL: NCT07252375
Title: A Single-Arm, Exploratory, Self-Controlled Clinical Study of Hetrombopag for Secondary Prevention of Thrombocytopenia Induced by Gemcitabine Plus Cisplatin in the Treatment of Nasopharyngeal Carcinoma
Brief Title: A Clinical Study of Hetrombopag for Prevention of Thrombocytopenia Induced by Gemcitabine Plus Cisplatin in the Treatment of Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HQBP01
Record Dates: First submitted 2025-11-16; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Nasopharyngeal Carcinoma (NPC); CTIT-Chemotherapy Induced Thrombocytopenia
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Secondary Prevention Cohort (Experimental)
  Interventions: Drug: herombopag olamine tablets

INTERVENTIONS:
Drug: herombopag olamine tablets — Oral Hetrombopag Olamine Tablets will be initiated at a daily dose of 5 mg (initial dose) on Day 1 (D1) of each chemotherapy cycle, and administered continuously until the start of the next chemotherapy cycle. During the oral administration period, blood routine examinations of subjects will be collected every 3-5 days, and the dosage of hetrombopag will be adjusted according to the Platelet Count (PIT). The dosage adjustment rules are as follows:
  When PLT ≥ 100 × 10⁹/L, discontinue administration; When 50 × 10⁹/L ≤ PLT < 100 × 10⁹/L, increase the daily dose by 2.5 mg; When PLT < 50 × 10⁹/L, increase the daily dose by 5 mg; Note: When the platelet count is < 10.0 × 10⁹/L or there is a bleeding risk, rescue measures such as platelet transfusion may be considered based on clinical practice.

SUMMARY:
This study is a single-arm, exploratory, self-controlled clinical trial for the prevention of thrombocytopenia induced by gemcitabine plus cisplatin in the treatment of nasopharyngeal carcinoma. It aims to investigate the efficacy and safety of hetrombopag for the secondary prevention of thrombocytopenia caused by gemcitabine plus cisplatin in patients with nasopharyngeal carcinoma. The study protocol has been reviewed and approved by the Institutional Ethics Committee of Fujian Cancer Hospital, allowing the conduct of this clinical study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 18 to 75 years old, regardless of gender;
* 2. Patients with nasopharyngeal carcinoma confirmed by pathological or cytological examination;
* 3. Currently receiving treatment with the Gemcitabine + Cisplatin (GP) regimen at a 21-day cycle, with the lowest platelet count < 75×10⁹/L in the previous chemotherapy cycle, and expected to maintain the same chemotherapy regimen for at least 2 more cycles;
* 4. Estimated survival time ≥ 12 weeks;
* 5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-2;
* 6. Laboratory test indicators meeting the following requirements:

  1. Absolute Neutrophil Count (ANC) > 1.0×10⁹/L, Hemoglobin (Hb) > 80 g/L;
  2. Renal function: Creatinine (Cr) ≤ 1.5 × Upper Limit of Normal (ULN) or estimated Glomerular Filtration Rate (eGFR) ≥ 60 ml/min (calculated by the Cockcroft-Gault formula);
  3. Liver function: Total Bilirubin (TBIL) ≤ 1.5 × ULN; Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 3 × ULN; (If the patient has intrahepatic cholangiocarcinoma or liver metastasis, total bilirubin ≤ 3 × ULN and transaminases ≤ 5 × ULN);
  4. Coagulation function: International Normalized Ratio (INR) of Prothrombin Time (PT) ≤ 1.5 × ULN, and Activated Partial Thromboplastin Time (APTT) within the normal range;
* 7. Females of childbearing potential must agree to use contraception during the study and for 6 months after the study ends; non-lactating females are eligible. Males must agree to use contraception during the study and for 6 months after the study ends;
* 8. No participation in other clinical trials of drugs within 4 weeks prior to enrollment;
* 9. Subjects must understand the study details and voluntarily sign the Informed Consent Form (ICF);
* 10. No severe complications such as active massive gastrointestinal bleeding, perforation, jaundice, gastrointestinal obstruction, or non-cancerous fever > 38℃;
* 11. Expected to have good compliance and be able to complete follow-up for efficacy and adverse reactions as required by the protocol.

Exclusion Criteria:

* 1. Thrombocytopenia not caused by cancer therapy occurring within 6 months prior to screening, including but not limited to hepatic cirrhosis with hypersplenism, infection, and bleeding;
* 2. Having other hematopoietic system diseases besides chemotherapy-induced thrombocytopenia, including leukemia, primary immune thrombocytopenia (ITP), myeloproliferative diseases (MPDs), multiple myeloma (MM), myelodysplastic syndromes (MDS), etc.;
* 3. Complicated with bone marrow involvement or bone marrow metastasis;
* 4. Having received pelvic, spinal radiotherapy or large-field bone irradiation within 3 months prior to screening;
* 5. History of any arterial or venous thrombosis occurring within 6 months prior to screening;
* 6. Clinical manifestations of severe bleeding (such as gastrointestinal bleeding) within 2 weeks prior to screening;
* 7. Severe cardiovascular diseases (e.g., NYHA Cardiac Function Classification Grade III-IV) within 6 months prior to screening, or patients with arrhythmias known to increase thromboembolic risk (such as atrial fibrillation [AF]), history of coronary artery stenting, angioplasty, or coronary artery bypass grafting (CABG);
* 8. Brain tumor or brain metastasis;
* 9. Having received platelet transfusion within 2 days prior to enrollment;
* 10. Having received treatment with recombinant human thrombopoietin (rhTPO), recombinant human interleukin-11 (rhIL-11), or thrombopoietin receptor agonist drugs (such as eltrombopag, avatrombopag) within 5 days prior to screening;
* 11. Patients with known or anticipated allergy or intolerance to the active ingredient or excipients of Hetrombopag Ethanolamine Tablets (excipients include: cellulose-lactose, low-substituted hydroxypropyl cellulose [L-HPC], magnesium stearate, film-coating premix);
* 12. Pregnant or lactating women;
* 13. Patients deemed ineligible for enrollment by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence Rate of Grade 3 or Higher Cancer Therapy-Induced Thrombocytopenia (CTIT) | From the initiation of oral drug administration to 30 days after the last dose of the oral drug

IPD SHARING:
Plan to Share IPD: No